CLINICAL TRIAL: NCT05695716
Title: Cardiovascular Systems, Inc. (CSI) Percutaneous Ventricular Assist Device (pVAD) Second in Human Study
Brief Title: CSI Percutaneous Ventricular Assist Device (pVAD) Second in Human Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled; termination was business decision after acquisition of CSI by Abbott.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLN-0017-P
Record Dates: First submitted 2023-01-10; First posted 2023-01-25 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
Keywords: PCI; pVAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, single-site study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CSI pVAD System (Experimental): clinical use of the CSI pVAD System during high risk percutaneous coronary interventions (HR-PCI)
  Interventions: Device: CSI pVAD System

INTERVENTIONS:
Device: CSI pVAD System — The CSI percutaneous ventricular assist device (pVAD) is being investigated as a temporary left ventricular system intended to support and/or provide hemodynamic stability during high-risk percutaneous coronary interventions.

SUMMARY:
The purpose of this study is to collect data on safety and device performance on the CSI pVAD System used to support hemodynamic stability during HR-PCIs to inform device design and finalization.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. In the investigator's opinion, the subject is capable of providing informed consent.
3. Subject has signed the Independent Ethics Committee (IEC) approved study Informed Consent Form (ICF) prior to any study related procedures
4. Subject has a life expectancy ≥1 year
5. Subject has a left ventricular ejection fraction (LVEF) ≥15% and ≤40%
6. Subject has a planned elective or urgent high risk percutaneous coronary intervention with hemodynamic support
7. Subject of child bearing potential has a negative pregnancy test result

Exclusion Criteria:

1. Subject has ST-Elevation Myocardial Infarction (STEMI) within 30 days prior to study procedure based on criteria in SCAI definition
2. Subject has NSTEMI with cardiac enzymes that are not trending downward within 30 days prior to study procedure
3. Subject with RV failure (defined as reduced RV function on imaging and evidence of increased CVP >18 mmHg)
4. Subject with history of cardiac arrest within 30 days prior to study procedure requiring cardiopulmonary resuscitation OR any history of cardiac arrest with impairment in mental status, cognition or any global or functional neurological deficit
5. Subject is in cardiogenic shock (defined as systolic BP <90 mmHg, cardiac index <2.1 and/or evidence of impaired end organ perfusion) that is not responsive to fluid infusion or requiring any inotropic or pressor support
6. Subject received any pressors or inotropes within 24 hours prior to the start of the study procedure
7. Subject has evidence of current or prior endocarditis
8. Subject with active myocarditis
9. Subject had a deep vein thrombosis (DVT) or pulmonary embolism (PE) within 6 months prior to study procedure
10. Subject had a stroke or TIA within 6 months prior to study procedure
11. Subject had previous CABG within 6 months prior to study procedure
12. Subject had coronary intervention within 30 days prior to study procedure
13. Subject has a coronary intervention planned within 30 days post procedure
14. Subject has presence of left ventricular (LV) mural thrombus
15. Subject has history of valve replacement or repair (e.g., MitraClipTM) including transcatheter edge to edge repair (TEER)
16. Subject has significant mitral valve disease (defined as mitral regurgitation greater than moderate, grade ≥2+ by echocardiogram (ECHO), mitral stenosis with MVA <1.5 cm2) or has evidence of structural damage to the chordae tendineae or valve
17. Subject has significant aortic valve disease (defined as aortic stenosis (valve area ≤1.5 cm2 or moderate or severe aortic regurgitation (grade ≥2+ by ECHO))
18. Subject with atrial fibrillation present at the time of enrollment or any time prior to RHC or CSI pVAD device placement
19. Subject has sustained tachycardia with heart rate over 120 BPM
20. Subject has sustained ventricular tachycardia either pre- or during intervention
21. Subject has severe pulmonary hypertension, defined as mean pulmonary artery pressure ≥40 mmHg
22. Subject has presence of an aneurysm or dissection along vascular delivery path including:

    1. Abdominal aortic aneurysm 4.0 cm or greater, OR
    2. Significant descending thoracic aortic aneurysm greater than 4.5 cm, OR
    3. Any dissection of the ascending, transverse, or descending aorta
23. Subject has severe peripheral vascular disease that will preclude the use of a 12Fr access sheath, which is required for the insertion of the CSI pVAD catheter
24. Subject has severe aortic tortuosity
25. Subject has severe aortic calcification that may preclude appropriate placement of the CSI pVAD device
26. Subject's vasculature will not tolerate a right heart catheterization (RHC)
27. Subject has chronic renal dysfunction defined by either:

    1. Serum creatinine ≥ 2.5 mg/dl AND/OR
    2. Requires hemodialysis
28. Subject has liver dysfunction with either:

    1. Elevation of liver enzymes and bilirubin levels to ≥ 3X ULN OR
    2. Internationalized Normalized Ratio (INR) ≥ 2 OR
    3. Lactate dehydrogenase (LDH) > 2.5X ULN
29. Subject has uncorrectable abnormal coagulation parameters defined as either:

    1. Platelet count ≤75,000 per μL OR
    2. INR ≥2.0 or
30. Subject has history of heparin induced thrombocytopenia
31. Subject has history of bleeding diathesis or known coagulopathy, any recent GU or GI bleed within 30 days prior to study procedure or will refuse blood transfusions
32. Subject has anemia (hemoglobin <10.0 g/dL) or polycythemia/hypovolemia (hemoglobin >16.5 g/dL)
33. Subject requires, or, in the clinical judgement of the investigators may need, long term support (>6 hours) with a commercially available mechanical circulatory support (MCS) device
34. Subject was on any mechanical cardiac support device at any time within 14 days prior to the study procedure.
35. Subject has an active systemic infection requiring oral or intravenous antibiotics, or elevated temperature or white blood cell count that may be due to infection
36. Subject has been diagnosed with COVID ≤10 days prior to study procedure or is excluded due to COVID based on institution or other (e.g., CDC) guidelines
37. Subject has an allergy or intolerance to ionic and nonionic contrast media, anticoagulants, or antiplatelet therapy drugs that cannot be adequately premedicated
38. Subject has an allergy or intolerance to CSI pVAD System components
39. Subject is pregnant
40. Subject is currently participating or plans to participate in another investigational drug- or device trial that may affect any of this study's endpoints
41. Subject has any other anatomical-, clinical-, social-, etc. characteristics that preclude the subject from being a candidate for the study
42. Subject has any contradiction listed in the current IFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
CSI pVAD System device placement/procedural success | Intraprocedural
  Delivery of the device to the correct anatomical position, successful operation and removal of the CSI pVAD system
Prevention of severe hypotension while on CSI pVAD device support | Intraprocedural
  Percentage of subjects who were free from severe hypotension while on CSI pVAD device support.
Major Device-Related Adverse Events | from Intraprocedure through study exit at 30 day follow up
  Percentage of subjects who were free from:
  * Access site complications, defined as complications requiring unplanned transfusion of packed red blood cells (1 unit or more) and/or percutaneous or surgical intervention
  * Bleeding (BARC category 3 or 5, and category 2 if serious criterion is met)
  * Cardiovascular death
  * Clinically significant myocardial infarction (MI), classified based on the SCAI and Fourth Universal definitions
  * Stroke (ischemic or hemorrhagic), classified based on symptoms on CT or MRI imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Chambers, MD, Study Director — Abbott Medical Devices
Locations (1):
- Tbilisi Heart & Vascular, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No